CLINICAL TRIAL: NCT04013009
Title: Laparotomy Closure Techniques: do Surgeons Follow the Latest Guidelines? Results of a Questionnaire.
Status: Completed | Type: Observational
Sponsor: VieCuri Medical Centre (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Arthur Bloemen, resident general surgery, VieCuri Medical Centre
Other Study IDs: 01
Record Dates: First submitted 2019-07-02; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Incisional Hernia; Laparotomy Closure Technique
Keywords: incisional hernia; prevention; laparotomy closure; quality improvement; survey; guideline
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Incisional hernias after laparotomy are associated with significant morbidity and increased costs. Research is focused on development of new techniques to prevent incisional hernia. Little is known about application of this evidence in daily practice. Therefore, a survey was performed among Dutch surgeons.

DETAILED DESCRIPTION:
Incisional hernias after laparotomy are associated with significant morbidity and increased costs. Research is focused on development of new techniques to prevent incisional hernia. Little is known about application of this evidence in daily practice. Therefore, a survey was performed among Dutch surgeons.

All members of the Dutch Surgical Society were invited to participate in a 24-question online survey on techniques and materials used for abdominal wall closure after midline laparotomy. Subgroup analysis based on surgical subspecialty, hospital and experience was performed.

ELIGIBILITY:
Inclusion Criteria:

* surgeon in the Netherlands

Exclusion Criteria:

* not practicing surgery
* not practicing in the Netherlands

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Surgeons in the Netherlands
Sampling Method: Non-Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
opinions on and current technique used for laparotomy closure | July till August 2016 at survey completion; snapshot measurement
  multiple choice questions
knowledge of incisional hernia development | July till August 2016 at survey completion; ; snapshot measurement
  multiple choice questions

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Bloemen, MD, Principal Investigator — VieCuri Medical Centre

IPD SHARING:
Plan to Share IPD: Undecided
anonymous individual data will be provided upon request